CLINICAL TRIAL: NCT06544434
Title: Laser Acupuncture for Meniere Disease: A Randomized Controlled Trial
Brief Title: Laser Acupuncture for Meniere Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAMD-RCT-2024
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Meniere Disease
Keywords: Meniere Disease; RCT; Laser acupuncture
MeSH Terms: conditions — Meniere Disease | interventions — Lasers; Betahistine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser acupuncture 3 month Group (Experimental)
  Interventions: Device: Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy); Drug: Betahistine Mesylate tablet
- Sham acupuncture Group (Sham Comparator)
  Interventions: Device: Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy); Drug: Betahistine Mesylate tablet
- Control Group (Other)
  Interventions: Drug: Betahistine Mesylate tablet

INTERVENTIONS:
Device: Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy) — MLS laser is a class IV NIR laser with two synchronized sources (905 nm with 75 W peak power, pulsed mode; 808 nm with power 1 W, continuous mode). Both laser beams were synchronized, the locked waves work with the range 1-2000 Hz.
  Arms: Laser acupuncture 3 month Group; Sham acupuncture Group
Drug: Betahistine Mesylate tablet — Betahistine Mesylate tablet (Merislon, Eisai Co., Ltd., China) with the treatment of 6 mg, 3 times a day.

SUMMARY:
Objective: To evaluate the effect of laser acupuncture for the patients Meniere disease.

Methods: We enrolled 324 patients at Beijing Tongren Hospital. Patients completed outcome measures at baseline, 3 months, 6 months, and 12 months. Video head impulse test (vHIT), The Caloric Test, Tinnitus Handicap Inventory (THI), Dizziness Handicap Inventory (DHI), Pure Tone Audiometry (PTA), and visual scale of ear stuffiness to evaluate the therapeutic effects. A difference of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of meniere disease.

Exclusion Criteria:

1. Serious mental illness or social problems, and neurological disorders, and systemic diseases, such as malignant tumors, and other serious consumptive diseases.
2. Planning for pregnancy, those in pregnancy, or those who were lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | Baseline, month 3, 6 and 12
  The DHI is 25-items self-reported questionnaire that used to evaluate the functional, emotional, and physical impact of dizziness on patients' daily life. Among the overall 25 items of questions, 9 items are emotional related, 9 items are functional related, and 7 items are physical related questions. The three answer options are "yes," "sometimes," and "no," with scores of 4, 2, and 0, respectively. The overall score is the sum of 25 items (Range: 0-100). Higher scores equate to greater severity of dizziness symptoms.
Tinnitus Handicap Inventory (THI) | Baseline, month 3, 6 and 12
  The THI is a 25-items, self-reported questionnaire regarding tinnitus handicap in daily life. The questionnaire comprises a 12-item functional subscale, an 8-item emotional subscale, and a 5-item catastrophic subscale. The three answer options are "yes," "sometimes," and "no," with scores of 4, 2, and 0, respectively. The overall score is the sum of 25 items (Range: 0-100). Higher scores equate to greater severity of tinnitus symptoms.
Pure tone thresholds (PTA) | Baseline, month 3, 6 and 12
  The pure tone thresholds was performed in a sound-attenuated, double-walled booth with circumaural headphones (Sennheiser HD 280 for frequencies from 250 to 8000 Hz and Sennheiser HD 200 for frequencies from 8000 to 14000 Hz; Sennheiser, Old Lyme, USA) on a certified and calibrated audiometric system (Interacoustics, Middelfart, Denmark). Thresholds were measured using a probe-detection paradigm with pure tones presented for 250 ms at frequencies of 250, 500, 1000, 2000, 4000, 8000 Hz for each ear. To determine the LDL, the volume was set to 75 dB at 1000 Hz and then continuously raised in 5 dB steps (every 5 s) until the subject gave the signal that this volume was uncomfortable.
  When the volume exceeded 110 dB the test was stopped to prevent any hearing damage.
  The severity of hearing impairment was calculated as mild (20-40 dB), moderate (41-70 dB), severe (71-95 dB) and profound (>95 dB). Normal hearing was defined as pure-tone thresholds less than 20 dB.
Visual analogue scale (VAS) | Baseline, month 3, 6 and 12
  The VAS scale of aural fullness consists of a 100 mm straight line with defined endpoints ("no aural fullness" and "worst aural fullness imaginable") on which the patients were asked to mark their experienced aural fullness (results in mm) at the actual time ("VAS now"). The higher VAS score (Range: 0-100) is correlated with a severe aural fullness.

SECONDARY OUTCOMES:
Video head impulse test (vHIT) | Baseline, month 3, 6 and 12
  vHIT was used to assess the function of all the six SCCs by measuring the gain of the vestibulo-ocular reflex. The instrument comprises an inertial measurement unit to measure movements of the head and an infrared camera to record eye movements. vHIT can calculate the mean gain value (ratio of eye to head velocity) for each of the six SCCs, and also detect covert or overt saccades. During the test, goggles were secured firmly to patients' head to ensure that the goggles did not slip from the face during head movement. Patients sat ~1.5 m in front of a wall on which a visual target was affixed. Before testing, head movement and eye movement were calibrated according to the manufacturer's instructions. According to manufacture recommendations, normal gain values are expected to range between 0.80 and 1.20 for horizontal canals, and 0.70-1.20 for vertical canals. Pathological saccades and gain values below the normal range were recorded.
The Caloric Test | Baseline, month 3, 6 and 12
  The caloric test was employed to evaluate the horizontal semicircular canal (SCC). The patients took supine position and raised their head to 30 degrees with a pillow. The right and left ears of the patients were stimulated with cool air (24°C) and warm air (50°C) by using an air caloric irrigator system (Micromedical Technologies Inc., Chatham, IL, USA) and a Brookler-Grams closed-loop irrigation unit. We used videonystagmography (VNG) (Ulmer Inc. Marseille, France) to record horizontal eye movements during the test. The subjects were perfused four times for 60 s.
  After perfusion, the nystagmus was observed for 60 s. Unilateral Weakness (UW) was calculated using the maximal slow phase eye velocity: UW = | (RC + RW) - (LC + LW) | / (RC + RW +LC + LW) × 100%, where RC = right cool, RW
  = right warm, LC = left cool, and LW = left warm. UW >25% was considered abnormal.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing TongRen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: From the study publication to 5 years
Access Criteria: email